# Non-Interventional Study (NIS) Protocol

| Document Number: | NA |
|---|---|
| BI Study Number: | 1199-0523 |
| Bl Investigational Product(s): | Not applicable |
| Title: | Incidence probability of progression to progressive fibrosing interstitial lung diseases and status of management and treatments in patients with fibrosing interstitial lung diseases other than idiopathic pulmonary fibrosis in Japan |
| Brief lay title: | Study of progression to PF-ILD incidence/management and treatment |
| Protocol version identifier: | 1.4 |
| Date of last version of protocol: | 29 Nov. 2023 |
| PASS: | Not applicable |
| EU PAS register number: | Not applicable |
| Active substance: | Not applicable |
| Medicinal product: | Not applicable |
| Product reference: | Not applicable |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | |
| Joint PASS: | Not applicable |
| Research question | PRIMARY OBJECTIVE |
| and objectives: | To investigate the incidence probability of progression to PF-ILDs in patients with fibrosing ILD other than IPF in real-world setting in Japan |
| | SECONDARY OBJECTIVE |
| | To investigate the characteristics of procedures for management and treatment in patients with fibrosing ILD other than IPF in real-world setting in Japan |
| Country(-ies) of study: | Japan |
| Author: | |
| Co-Author: | |

| Marketing authorisation holder(s): | |
|-------------------------------------------|----------------|
| In case of PASS, add: MAH contact person: | Not applicable |
| In case of PASS, add: | Not applicable |
| In case of PASS, add: | Not applicable |
| Date: | 29 Nov. 2023 |
| | Page 1 of 41 |

# Proprietary confidential information

© 2024 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

## 1. TABLE OF CONTENTS

| 1. | TABLE OF CONTENTS | 3 |
|---|---|---|
| 2. | LIST OF ABBREVIATIONS | 4 |
| 3. | RESPONSIBLE PARTIES | 5 |
| 4. | ABSTRACT | 5 |
| 5. | AMENDMENTS AND UPDATES | 8 |
| 6. | MILESTONES | 9 |
| 7. | RATIONALE AND BACKGROUND | 10 |
| 8. | RESEARCH QUESTION AND OBJECTIVES | 11 |
| 8.1 | PriMary Objective | 11 |
| 8.2 | Secondary objective | 11 |
| 9. | RESEARCH METHODS | |
| 9.1 | STUDY DESIGN | 11 |
| 9.2 | SETTING | 11 |
| 9.3 | VARIABLES | 13 |
| 9.4 | DATA SOURCES | 15 |
| 9.5 | STUDY SIZE | 15 |
| 9.6 | DATA MANAGEMENT | 15 |
| 9.7 | DATA ANALYSIS | 15 |
| 9.8 | QUALITY CONTROL | 17 |
| 9.9 | | |
| 9.1 | 0 OTHER ASPECTS | 17 |
| 10. | PROTECTION OF HUMAN SUBJECTS | 17 |
| 11. | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 17 |
| 12 | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| | REFERENCES | |
| | 1 PUBLISHED REFERENCES | |
| | 2 UNPUBLISHED REFERENCES | |
| | EX 1. LIST OF STAND-ALONE DOCUMENTS | |
| | EX 2. INTERSTITIAL LUNG DISEASE PROGRESSION PROXIES | |
| | EX 3. Code for Treatment, Management & clnical examination | |
| | EX 4. Code for Comorbidity and medical history | |
| | EX 5. ALGORITHMS FOR DEFINING uderlying diseases | |
| | EX 6. Information of the code to define fibrosing ILD and underlying diseases | |
| | EX 7 REVIEWERS AND APPROVAL SIGNATURES | ۰۰۰ ۲ |

#### 2. LIST OF ABBREVIATIONS

COPD Chronic Obstructive Pulmonary Disease

CTD-ILD Connective Tissue Disease-Interstitial Lung Disease

DPC Diagnosis Procedure Combination
HP Hypersensitivity Pneumonitis

HRCT/CT High-Resolution Computed Tomography/Computed Tomography

ILD Interstitial Lung Disease IHD Instant Health Data

IIPs Idiopathic Interstitial Pneumonias

iNSIP Idiopathic Nonspecific Interstitial Pneumonia

IPF Idiopathic Pulmonary Fibrosis KL-6 Krebs von den Lungen-6

MCTD Mixed Connective Tissue disease

MDV Medical Data Vision

PF-ILD Progressive Fibrosing Interstitial Lung Disease

PM/DM-ILD Polymyositis/Dermatomyositis-Interstitial Lung Disease

RA-ILD Rheumatoid Arthritis-Interstitial Lung Disease

SAS Statistical Analysis System

SLE-ILD Systemic Lupus Erythematosus-Interstitial Lung Disease

SP-D Surfactant Protein D

SSc-ILD Systemic Sclerosis-Interstitial Lung Disease

| 3. | RESPONSIBLE PARTIES |
|----------|-----------------------------------|
| NIS | |
| Co-NIS | |
| Data Mar | nagement and Statistical Analysis |
| Medical | Advisor |
| Data sou | irce |

## 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim Co., Ltd. | | | |
| Name of finish product: Not applica | ed medicinal | | |
| Name of active ingr | edient: | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| DD Month YYYY | | 1.4 | 29 Nov. 2023 |
| Title of study: | Incidence probability of progression to progressive fibrosing interstitial lung diseases and status of management and treatments in patients with fibrosing interstitial lung diseases other than idiopathic pulmonary fibrosis in Japan | | |
| Rationale and background: | While idiopathic pulmonary fibrosis (IPF) is the best-known progressive fibrosing interstitial lung disease (PF-ILD), there is a group of patients with different underlying clinical interstitial lung disease (ILD) diagnoses other than IPF who develop a progressive fibrosing phenotype during the course of their disease. There is minimal literature available to estimate the proportion of patients | | |
| | who develop PF-ILDs in patients with fibrosing ILD other than IPF and, the current management and treatment for these diseases are not well-known in Japan. These information are keys to gaining a better understanding of the size of | | |
| | this population with high unmet need and for physicians, patients and other stakeholders to optimize allocation of resources, diagnostic assessment and management of this patient population. | | |
| Research | PRIMARY OBJE | CTIVE | |
| question and objectives: | To investigate the incidence probability of progression to PF-ILDs in patients with fibrosing ILD other than IPF in real-world setting in Japan SECONDARY OBJECTIVE | | |
| | To investigate the characteristics of procedures for management and treatment in patients with fibrosing ILD other than IPF in real-world setting in Japan | | |
| Study design: | This is a retrospective cohort study using the database from Medical Data Vision (MDV). | | |
| | that each patient<br>encounter in the<br>in the period from<br>patient who mee<br>will be followed<br>period (i.e., 28- | n-2012 to 28-May-2020 will be to it is observable from his/her fit database. The patients with fit om 01-Jan-2013 to 6 months at all the inclusion criteria and up from the day after the inde May-2020), the last encounted whichever occurs first. | irst encounter to his/her last<br>brosing ILD will be identified<br>before 28-May-2020. Each<br>none of the exclusion criteria<br>x date until the end of study |

| Population: | Patients who meet all of the inclusion criteria and do not meet any of the exclusion criteria will be included in the study population. |
|---|---|
| | Inclusion Criteria: |
| | <ol> <li>Patients diagnosed with at least two fibrosing ILD codes on different<br/>dates in the patient identification period from 01-Jan-2013 to 6<br/>months before 28-May-2020</li> </ol> |
| | Patients aged 18 years and older on the index date |
| | <ol> <li>Patients for whom data for the 12 months prior to the index date can<br/>be extracted as baseline data</li> </ol> |
| | Exclusion Criteria: |
| | <ol> <li>Patients grouped into the underlying disease of IPF</li> <li>Patients who have met PF-ILD progression criteria during the baseline period</li> </ol> |
| | Note: only diagnosis records without 'suspect flag' are to be considered for evaluating diagnosis related in/excl criteria" |
| Variables: | The following information will be extracted from MDV database in this study; sex, age, comorbidity and medical history of interest, Underlying disease (pre-specified ILD), clinical examination, treatment and management of interest |
| Data sources: | The MDV database consists of anonymized administrative claims and Diagnosis Procedure Combination (DPC) data for inpatient and outpatient settings from acute hospitals (mainly considered as advanced treatment hospitals). The database includes >35 million patients from >400 hospitals. |
| | Patients in Japan have free access to health care facilities and data from the other hospitals not included in the database are unavailable. |
| Study size: | The planned sample size is not based on the formal statistical hypothesis testing and statistical precision. Because the MDV database consists of >35 million patients, it is expected that the sufficient number of non-IPF fibrosing ILD patients will be included in the study. |
| Data analysis: | Primary outcome Incidence probability of progression to PF-ILDs at 6, 12, 18, and 24 months after the index date. |
| | Cumulative incidence probability will be estimated by using Kaplan-Meier method. |
| | Secondary outcomes |
| | Management and treatment during follow-up period |
| | Frequency of patients with management and treatment of interest during follow-up period will be analyzed descriptively. |
| Milestones: | - Final protocol: 28 Mar 2023 |
| | - IRB approval: Prior to study start |
| | - Start of data analysis: After the IRB approval |
| | - Final results: Q2 2023 |
| | - Final study report: Q3 2023 |
| | - Publications: Q3, 2023 |

# 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | 28 March 2023 | 9.2.2.1<br>Exclusion<br>Criteria | 2)Patients who have met PF-ILD progression criteria during the baseline period and 3) delete | To further clarify<br>and simplify the<br>exclusion criteria |
| 2 | 21 Sep. 2023 | ANNEX 2 and 3 | Add Generic<br>names and<br>correct ATC<br>codes | To correct the drug codes |
| 3 | 21 Sep. 2023 | ANNEX 2 and 3 | *transdermal patch, sublingual agent, Transmucosal agent, suppository are excluded | To reflect the updated definition of opioid use |
| 4 | 10 Nov. 2023 | ANNEX 2 and 3 | K514-4<br>K514-6 | To correct codes for<br>lung transplant |
| 5 | 29 Nov. 2023 | ANNEX 2 and 3 | N02A0 | To correct the drug code for opioid |

# 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------|------------------------|
| IRB/IEC approval | Prior to study start |
| Start of Data Analysis | After the IRB approval |
| Interim Report | NA |
| Final report of study results: | Q3 2023 |

#### 7. RATIONALE AND BACKGROUND

The term interstitial lung disease (ILD) encompasses a large group of over 200 pulmonary disorders. While idiopathic pulmonary fibrosis (IPF) is the best-known progressive fibrosing ILD (PF-ILD), there is a group of patients with different underlying clinical ILD diagnoses other than IPF who develop a progressive fibrosing phenotype during the course of their disease (e.g., idiopathic interstitial pneumonias [IIPs] such as idiopathic nonspecific interstitial pneumonia [iNSIP] and unclassifiable IIP; hypersensitivity pneumonitis [HP]; autoimmune interstitial lung disease [connective tissue disease-ILDs (CTD-ILD) such as rheumatoid arthritis-ILD (RA-ILD), systemic sclerosis-ILD (SSc-ILD) and anti-synthetase syndrome]; Sarcoidosis; Pneumoconiosis/exposure related ILD) [P17-10582, P18-04729, P19-01738, R19-0854]. These patients demonstrate a number of similarities to patients with IPF, with their disease being defined by the presence of progressive pulmonary fibrosis, worsening respiratory symptoms, declining lung function despite immunomodulatory therapies and, ultimately, early mortality.

Although there had been no indicated therapies for patients with chronic fibrosing ILDs with a progressive phenotype (other than IPF), Nintedanib has just been approved for SSc-ILD in the end of Dec. 2019 based on the results of the SENSCIS trial (NCT02597933) [P19-04387] and for PF-ILDs in the end of May 2020 in Japan based on the results of the INBUILD trial (NCT02999178) [P19-08802, P20-02333].

There is minimal literature available to estimate the proportion of patients who develop PF-ILDs in patients with fibrosing ILD other than IPF in Japan. In addition, the current management and treatment for these diseases are not well-known. These information are keys to gaining a better understanding of the size of this population with high unmet need and for physicians, patients and other stakeholders to optimize allocation of resources, diagnostic assessment and management of this patient population.

Therefore, this study will use the database from Medical Data Vision (MDV) to investigate the incidence probability of progression to PF-ILDs according to each co-existing underlying diseases and the characteristics of procedures for management and treatment in patients with fibrosing ILD other than IPF.

#### 8. RESEARCH QUESTION AND OBJECTIVES

#### 8.1 PRIMARY OBJECTIVE

To investigate the incidence probability of progression to PF-ILDs in patients with fibrosing ILD other than IPF in real-world setting in Japan

#### 8.2 SECONDARY OBJECTIVE

To investigate the characteristics of procedures for management and treatment in patients with fibrosing ILD other than IPF in real-world setting in Japan

#### RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a retrospective cohort study using the database from MDV.

Data from 01-Jan-2012 to 28-May-2020 will be used. It will be considered that each patient is observable from his/her first encounter to his/her last encounter in the database. The patients with fibrosing ILD will be identified in the period from 01-Jan-2013 to 6 months before 28-May-2020. Each patient who meets all the inclusion criteria and none of the exclusion criteria will be followed up from the day after the index date\* until the end of study period (i.e. 28-May-2020), the last encounter in the MDV database, in-hospital death, whichever occurs first.

\*The index date will be the date of the second diagnosis of fibrosing ILD. Please refer to the Section 9.2.2.1 for the detailed codes of fibrosing ILD.



 $<sup>^{\</sup>star}$ The index date will depend on the time the patient fulfils the eligibility criteria

Figure 1 . Schematic of the Study Design

#### 9.2 SETTING

#### 9.2.1 Study sites

There are no study sites for this study because it is a database study.

#### 9.2.2 Study population

#### 9.2.2.1 Eligibility criteria

Patients who meet all of the inclusion criteria and do not meet any of the exclusion criteria will be included in the study population.

#### **Inclusion Criteria:**

- 1) Patients diagnosed with at least two fibrosing ILD codes\*1 on different dates in the patient identification period from 01-Jan-2013 to 6 months before 28-May-2020
- 2) Patients aged 18 years and older on the index date
- 3) Patients for whom data for the 12 months prior to the index date can be extracted as baseline data
  - \*1 International Statistical Classification of Diseases and Related Health Problems (ICD-10) code or disease code: J84.1, J84.9, 8844510, 8848382, 8844341, 8848278, 8836513, 8848267, 8848302, 8839362, 8848283, 8837013, 8834158, 8848245, 8840951, 8847737

#### **Exclusion Criteria:**

- 1) Patients grouped into the underlying disease of IPF\*1
- 2) Patients who have met PF-ILD progression criteria during the baseline period
  - \*1 Please refer to the ANNEX 5 for algorithm to define underlying diseases

Note: only diagnosis records without 'suspect flag' are to be considered for evaluating diagnosis related in/excl criteria"

#### 9.3 VARIABLES

#### 9.3.1 Outcomes

#### 9.3.1.1 Primary outcome

Incidence probability of progression to PF-ILDs at 6, 12, 18, and 24 months after the index date\*

Progression to PF-ILD as event in this study is defined in Table 1 as well as Annex 2. Event date will be the date when the one of criteria of the progression to PF-ILD is met.

\*The index date will be the date of the second diagnosis of fibrosing ILD. Please refer to the Section 9.2.2.1 for the detailed codes of fibrosing ILD.

Table 1. Interstitial lung disease progression proxies

#### Proxv

- ≥ 3 pulmonary function tests on different dates of service within 365 days
- The date of the 3<sup>rd</sup> pulmonary function test will be the date of progression
- ≥ 3 HRCT/CT on different dates of service within 365 days
- The date of the 3rd HRCT/CT will be the date of progression
- ≥ 1 claim for oxygen therapy (HOT) during follow-up period
- ≥ 1 respiratory hospitalization during follow-up period
- ≥ 1 claim for palliative care during follow-up period
- ≥ 1 lung transplant during follow-up period
- ≥ 1 new\* claim for immunosuppressive drugs during follow-up period with at least two out of the three test codes\*\* within 3 months before new claims for immunosuppressive drugs

Rituximab

**Tacrolimus** 

Mycophenolate

Cyclosporine

Cyclophosphamide

Azathioprine

**Tocilizumab** 

- \*: Not received in the 12 months prior to the index date
- \*\*: 1) Pulmonary function tests, 2) HRCT/CT, 3) KL-6 or SP-D
- ≥ 1 new\* claim for oral corticosteroid with a prednisone-equivalent dose of >20 mg during follow-up period and with at least two out of the three test codes\* within 3 months before new claims for oral corticosteroid
- \*: Not received in the 12 months prior to the index date
- \*\*: ① Pulmonary function tests, ② HRCT/CT, ③ KL-6 or SP-D
- ≥ 1 claim for Nintedanib\* during follow-up period
- \*: Patients meeting this criterion will be counted only if patients with fibrosing ILDs meet this criterion on or after 29-May-2020, because nintedanib was approved for PF-ILD on 29-May-2020. Even if patients with fibrosing ILDs meet this criterion on or before 28-May-2020, they will not be counted.

HRCT; high-resolution computed tomography, CT; computed tomography, KL-6; krebs von den lungen-6, SP-D; surfactant protein D

#### 9.3.1.2 Secondary outcome

Management and treatment during follow-up period

The management and treatment of interest are shown in **Table 2**.

## 9.3.2 Covariates

The following information will be extracted from MDV in this study.

Table 2. Definition of variables

| Age Inde<br>Comorbidity and 12 | dex date dex date months before the te (included) | | Male/Female Age at Index date - Coronary heart disease - Gastro-esophageal reflux disease - Obstructive sleep apnoea syndrome - Chronic obstructive pulmonary disease (COPD) |
|---|---|---|---|
| Comorbidity and 12 | months before the | | - Coronary heart disease - Gastro-esophageal reflux disease - Obstructive sleep apnoea syndrome |
| | | index | <ul><li>Gastro-esophageal reflux disease</li><li>Obstructive sleep apnoea syndrome</li></ul> |
| medical history date | te (included) | | - Obstructive sleep apnoea syndrome |
| | | | - Chronic obstructive pulmonary disease (COPD) |
| | | | - Lung cancer |
| | | | - Pulmonary hypertension |
| 1 | | | See Annex 4 for code to define each comorbidity and |
| | | | medical history |
| , , | months before the | index | , , |
| AND THE RESIDENCE OF THE PARTY | te (included) | | Non-autoimmune ILD, Multiple, Unknown) |
| (Pre-specified ILD) | | | <ul> <li>ILD Category (Hypersensitive pneumonitis, Exposure-<br/>related ILD, idiopathic nonspecific interstitial<br/>pneumonia (iNSIP), Unclassifiable idiopathic<br/>interstitial pneumonias (IIP), Sarcoidosis, RA-ILD, SSc-<br/>ILD, mixed connective tissue disease-ILD (MCTD-ILD),<br/>Other autoimmune ILD, Other ILD, Multiple, Unknown)</li> </ul> |
| | | | <ul> <li>Pre-Specified ILD Clinical Diagnosis (Hypersensitive<br/>pneumonitis, Exposure-related ILD, iNSIP,<br/>Unclassifiable IIP, Sarcoidosis, RA-ILD, SSc-ILD,<br/>MCTD-ILD, Systemic Lupus Erythematosus-ILD (SLE-ILD), Polymyositis/Dermatomyositis-ILD (PM/DM-ILD),<br/>Sjogren ILD, Other autoimmune ILD, Other ILD,<br/>Multiple, Unknown)</li> </ul> |
| | | | See Annex 5 for algorithm to define underlying diseases |
| A CONTRACTOR OF THE PROPERTY O | months before the | index | - Rituximab |
| date | te (included) | | - Tacrolimus |
| - | | | - Mycophenolate |
| Foll | llow-up period | | - Cyclosporine |
| | | | - Cyclophosphamide |
| | | | - Azathioprine |
| | | | - Oral Corticosteroid |
| | | | - Tocilizumab |
| | | | - Nintedanib |
| | | | See Annex 3 for code to define each treatment |
| | | | As for corticosteroid and immunosuppressive drugs during follow-up period, the same condition used for criteria of progression to PF-ILD will be applied. |
| Management Foll | llow-up period | | - Oxygen therapy (HOT) |
| | | | - Lung transplant |
| | | | - Palliative care (oxygen inhalation, opioid use) |
| | | | See Annex 3 for code to define each management |
| | months before the | index | - Pulmonary function test |
| examination date | te (included) | | - HRCT/CT |
| | | | - KL-6 |
| | | | - SP-D |
| | | | See Annex 3 for code to define each clinical examination |

#### 9.4 DATA SOURCES

The MDV database consists of anonymized administrative claims and DPC data for inpatient and outpatient settings from acute hospitals (mainly considered as advanced treatment hospitals). At present, the database includes >35 million patients from >400 hospitals. Patients in Japan have free access to health care facilities and data from the other hospitals

not included in the database are unavailable.

#### 9.5 STUDY SIZE

The planned sample size is not based on the formal statistical hypothesis testing and statistical precision. Because the MDV database consists of >35 million patients, it is expected that the sufficient number of non-IPF fibrosing ILD patients will be included in the study.

#### 9.6 DATA MANAGEMENT

The anonymised data received from hospitals has been checked by data managers in MDV to update the database. The database Boehringer Ingelheim (BI) received from MDV will be used.

The analyses will be performed using Instant Health Data (IHD) platform, SAS statistical software (version 9.3 or higher) and/or R.

#### 9.7 DATA ANALYSIS

#### 9.7.1 Common handling for statistical analysis

Unless otherwise specified, descriptive analysis is planned.

The summary statistics for continuous variables are N, mean, standard deviation, minimum, 25<sup>th</sup> percentile (Q1), median, 75<sup>th</sup> percentile (Q3), and maximum.

Tabulations of frequencies for categorical variables will include all possible categories and will display the number of observations in a category as well as percentage (%) relative to the population analysed. The precision for percentage will be one decimal point.

#### 9.7.2 Statistical analysis

#### 9.7.2.1 Patient background characteristics and treatment

- Patient demographics (sex, age at the index date)
- Comorbidity and medical history during 12 months prior to the index date (included)
- Clinical examination, management, and treatment during 6 months prior to the index date (included)
- Duration of follow-up period, which is defined as "end of follow-up period" "start of follow-up period" + 1 day
- Underlying diseases

These will also be analysed in patients with progression to PF-ILD and those without progression to PF-ILD respectively.

#### 9.7.2.2 Primary outcome

- Incidence probability of progression to PF-ILDs at 6, 12, 18, and 24 months after the index date

Cumulative incidence probability of progression to PF-ILD at 6, 12, 18 and 24 months after the index date will be estimated by using Kaplan-Meier method. Greenwood's variance estimate will be used for calculating 95% confidence interval. Kaplan-Meier curve will also be displayed.

Of the patients with progression to PF-ILD, frequency of patients meeting each criteria of progression to PF-ILD will be analysed descriptively.

#### 9.7.2.3 Secondary outcomes

- Management and treatment during follow-up period Frequency of patients with management and treatment during follow-up period will be analyzed.

#### 9.7.3 Subgroup analysis

The three subgroup analyses by underlying diseases defined by disease codes on the index date and 12-months lookback period as described in Annex 5 will be performed for patient background characteristics and treatment, primary outcome, and secondary outcomes.

#### <Subgroup Patterns>

Underlying Autoimmune Disease (Subgroup1): Autoimmune ILD, Non-autoimmune ILD, Multiple, Unknown

ILD Category (Subgroup 2): Hypersensitive pneumonitis, Exposure-related ILD, iNSIP, Unclassifiable IIP, Sarcoidosis, RA-ILD, SSc-ILD, MCTD-ILD, Other autoimmune ILD, Other ILD, Multiple, Unknown

Pre-Specified ILD Clinical Diagnosis (Subgroup 3): Hypersensitive pneumonitis, Exposure-related ILD, iNSIP, Unclassifiable IIP, Sarcoidosis, RA-ILD, SSc-ILD, MCTD-ILD, SLE-ILD, PM/DM-ILD, Sjogren ILD, Other autoimmune ILD, Other ILD, Multiple, Unknown

#### 9.7.4 Sensitivity analysis

- 1) The end of data extraction period will be changed from 28-May-2020 to the latest data cut off. OFEV was approved for PF-ILD on 29-May-2020, and the characteristics of claims data before and after the above approval for new indications might not be different. To increase the sample size, all the analyses will be repeated with this data extraction period.
- 2) The index date will be changed from the date of the second code of fibrosing ILD to the date of the first code of fibrosing ILD because there might be patients who are asked to visit hospitals annually after the first diagnosis. All the analyses will be repeated with this index date.

In addition, all the analyses will be repeated with both data extraction period and index date changed.

After exploring the proxy patterns among patients meeting the criteria of progression to PF-ILD as described in Section 9.7.2.2, a sensitivity analysis with modified progression criteria might be performed.

#### 9.8 QUALITY CONTROL

The analysis program and the data codes used in the analysis will be checked by someone different from the creator.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

The MDV database does not have pulmonary function test results and there have been no evidence on the validated algorithm to define fibrosing ILD patients other than IPF and progression to PF-ILD as events by using claims data. Therefore, the estimated incidence in this study might be biased and the sensitivity analysis by using different algorithm is planned to assess the robustness of the results.

Due to the characteristics of health care system in Japan as described in Section 9.4, data generated in the clinics/hospitals other than hospitals included in the MDV database are not captured and the incidence probability and frequency might be underestimated.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees. The quality assurance auditor will have access to all study-related files.

#### 9.10.2 Study records

Not applicable. (This study will not use Case Report Forms.)

#### 9.10.3 Completion of study

Not applicable.

#### 9.10.4 Protocol deviations

Deviations from the research protocol that may occur in this study include deviations from the procedures for handling databases and methods of analysis and reporting. Any deviations should be reported to the principal investigator by the co-investigator or contract research organization.

#### 9.10.5 Compensation available to the patient in the event of study related injury

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

The MDV data used in this study is existing information and does not involve the acquisition of new information. In addition, it is anonymized processed information and cannot identify individuals. Therefore, the protection of subjects does not apply to this study.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Not applicable based on secondary use of data without any potential that any employee of BI or agent working on behalf of BI will access individually identifiable patient data.

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results of this research will be presented at conferences and published in peer-reviewed journals.

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

- P17-10582 Flaherty KR, Brown KK, Wells AU, et al Design of the PF-ILD trial: a double-blind, randomised, placebo-controlled phase III trial of nintedanib in patients with progressive fibrosing interstitial lung disease BMJ Open Respiratory Research 2017;4:e000212. doi: 10.1136/bmjresp-2017-000212
- P18-04729 Wells AU, Brown KK, Flaherty KR, Kolb M, Thannickal Victor J. What's in a name? That which we call IPF, by any other name would act the same. European Respiratory Journal. 2018;51(5). Prevalence and characteristics of progressive fibrosing interstitial lung disease in a prospective registry
- R11-4318 Guidelines for Good Pharmacoepidemiology Practices (GPP) (revision 2: April 2007). http://www.pharmacoepi.org/resources/guidelines\_08027.cfm (access date: 13 September 2011); Bethesda: International Society for Pharmacoepidemiology (ISPE) (2007)
- R15-4859 Guidance for industry and FDA staff: best practices for conducting and reporting pharmacoepidemiologic safety studies using electronic healthcare data (May 2013, drug safety). http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformati on/guida nces/ucm243537.pdf (access date: 28 August 2015); U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER) (2013)
- R15-48701 European Medicines Agency (EMA). The ENCePP code of conduct for independence and transparency in scientific the conduct pharmacoepidemiological and pharmacovigilance studies (London, EMA/929209/2011). November 2011. http://www.encepp.eu/code of conduct/documents/CodeofConduct Rev2.pd f (access date: 28 August 2015); London: European Medicines Agency (EMA), for Pharmacoepidemiology European Network of Centres Pharmacovigilance (ENCePP) (2011)
- P19-01738 Cottin V, Wollin L, Fischer A, Quaresma M, Stowasser S, Harari S. Fibrosing interstitial lung diseases: knowns and unknowns. Eur Resp Rev 2019;28:180100.
- R19-0854 Kolb M, Vasakova M. The natural history of progressive fibrosing interstitial lung diseases. Respir Res (Lond) 2019;20(1):57
- P19-08802 Flaherty KR, Wells AU, Cottin V, Devaraj A, Walsh SLF, Inoue Y, et al, INBUILD Trial Investigators. Nintedanib in progressive fibrosing interstitial lung diseases. New England Journal of Medicine, published on September 29, 2019, doi: 10.1056/NEJMoa1908681; 2019, p. 1718-1727.
- P20-02333 Wells AU, Flaherty KR, Brown KK, Inoue Y, Devaraj A, Richeldi L, et al, INBUILD Trial Investigators. Nintedanib in patients with progressive fibrosing interstitial lung diseases subgroup analyses by interstitial lung disease diagnosis in the INBUILD trial: a randomised, double-blind, placebo-controlled, parallel-group trial. Lancet Respiratory Medicine, Published Online March 5, 2020, doi: 10.1016/S2213-2600(20)30036-9; 2020. p. 453-460.

## 13.2 UNPUBLISHED REFERENCES

None.

# **ANNEX 1. LIST OF STAND-ALONE DOCUMENTS**

| Number | Document<br>Reference Number | Date | Title |
|---|---|---|---|
| 1 | Annex 1 | 20 February 2023 | List of stand-alone documents |
| 2 | Annex 2 | 20 February 2023 | INTERSTITIAL LUNG DISEASE PROGRESSION PROXIES |
| 3 | Annex 3 | 20 February 2023 | CODE FOR TREATMENT,<br>MANAGEMENT & CLNICAL<br>EXAMINATION |
| 4 | Annex 4 | 20 February 2023 | CODE FOR COMORBIDITY<br>AND MEDICAL HISTORY |
| 5 | Annex 5 | 20 February 2023 | ALGORITHMS FOR DEFINING UDERLYING DISEASES |
| 6 | Annex 6 | 20 February 2023 | INFORMATION OF THE CODE<br>TO DEFINE FIBROSING ILD<br>AND UNDERLYING DISEASES |
| 7 | Annex 7 | 20 February 2023 | REVIEWERS AND APPROVAL SIGNATURES |

# ANNEX 2. INTERSTITIAL LUNG DISEASE PROGRESSION PROXIES

| | billing code / generic |
|---|---|
| Proxy | names / EphMRA ATC |
| | code |
| ≥ 3 pulmonary function tests on different dates of service within 365 | |
| days | 160062610 |
| | 160062710 |
| The date of the 3 <sup>rd</sup> pulmonary function test will be the date of | 160062810 |
| progression | |
| | 170022290 |
| | 170011710 |
| | 170011810 |
| | 170028610 |
| ≥ 3 HRCT/CT on different dates of service within 365 days | 170033410 |
| | 170034910 |
| The date of the 3rd HRCT/CT will be the date of progression | 170040210 |
| | 170040410 |
| | 170040610 |
| | 170040810 |
| | 170041010 |
| ≥ 1 claim for oxygen therapy (HOT) during follow-up period | 114003710 |
| = 1 stanti for oxygen therapy (1101) during follow-up period | |
| | A221 |
| | A379 |
| | A370 |
| | B250 |
| | B440 |
| | J00 |
| | J01.x |
| | J02.x |
| | J03.x |
| | J04.x |
| | J05.x |
| | J06.x |
| | J110 |
| | J12.x |
| | J13 |
| | J14 |
| | J15.x |
| | J160 |
| ≥ 1 respiratory hospitalization during follow-up period | J18.x |
| = 1 respirately respiration during relies appeared | J20x |
| | J21.x |
| | J22 |
| | J40 |
| | J41.x |
| | J42 |
| | J43.x |
| | J44.x |
| | J45.x |
| | J84.x |
| | J96.x |
| | Segment of disease based |
| | on DPC is "01: Disease |
| | name which input the most |
| | medical resources", "11: |
| | Main disease name", or |
| | "21: Disease name behind |
| | hospitalization" |
| | Oxygen inhalation: |
| ≥ 1 claim for palliative care during follow-up period | 140005610 |
| = 1 Statist for pullidate during follow-up period | |
| | Opioid use: |

| | N02A0 [Excluding methadone, buprenorphine, naloxonecombinations (Suboxone)] * *transdermal patch, sublingual agent, Transmucosal agent, suppository are excluded |
|---|---|
| ≥ 1 lung transplant during follow-up period | K514-4<br>K514-6 |
| ≥ 1 new* claim for immunosuppressive drugs during follow-up period with at least two out of the three test codes** within 3 months before new claims for immunosuppressive drugs Rituximab Tacrolimus Mycophenolate Cyclosporine Cyclophosphamide Azathioprine Tocilizumab *: Not received in the 12 months prior to the index date **: ① Pulmonary function tests, ② HRCT/CT, ③ KL-6 or SP-D ≥ 1 new* claim for oral corticosteroid with a prednisone-equivalent dose of >20 mg during follow-up period and with at least two out of | Rituximab/ L01G1 Tacrolimus/ L04X0 Mycophenolate/ L04X0 Cyclosporine or (Ciclosporin, Cyclosporin) / L04X0 Cyclophosphamide/ L01A0 Azathioprine/ L04X0 Tocilizumab/ M01C0 & L04C0 (Generic names/ MphMRA ATC codes which each drug is under) |
| the three test codes* within 3 months before new claims for oral corticosteroid *: Not received in the 12 months prior to the index date **: ① Pulmonary function tests, ② HRCT/CT, ③ KL-6 or SP-D | H02A2 excluding Florinef |
| ≥ 1 claim for Nintedanib* during follow-up period *: Patients meeting this criterion will be counted only if patients with fibrosing ILDs meet this criterion on or after 29-May-2020, because nintedanib was approved for PF-ILD on 29-May-2020. Even if patients with fibrosing ILDs meet this criterion on or before 28-May-2020, they will not be counted. | Nintedanib/ L01H9 & R07D0 (Generic name/ MphMRA ATC codes which nintedanib is under) |

# ANNEX 3. CODE FOR TREATMENT, MANAGEMENT & CLNICAL EXAMINATION

| Drug name / | Generic names/ Codes |
|---|---|
| Treatment Rituximab | Rituximab/ L01G1 |
| Tacrolimus | Tacrolimus/ L04X0 |
| Mycophenolate | Mycophenolate/ L04X0 |
| Cyclosporine | Cyclosporine or (Ciclosporin, Cyclosporin)/ L04X0 |
| Cyclophosphamide | Cyclophosphamide/ L01A0 |
| Azathioprine | Azathioprine/ L04X0 |
| Oral Corticosteroid | H02A2 excluding Florinef |
| Tocilizumab | Tocilizumab/ M01C0 & L04C0 |
| Nintedanib | Nintedanib/ L01H9 & R07D0 |
| Oxgen therapy (HOT) | 114003710 |
| Lung transplant | K514-4<br>K514-6 |
| Palliative care | Oxygen inhalation: 140005610 |
| | Opioid use: N02A0 [Excluding methadone, buprenorphine, naloxonecombinations (Suboxone)] * *transdermal patch, sublingual agent, Transmucosal agent, suppository are excluded |
| PFT | 160062610<br>160062710<br>160062810 |
| HRCT/CT | 170022290<br>170011710<br>170011810<br>170028610<br>170033410<br>170034910<br>170040210<br>170040410<br>170040610<br>170040810<br>170041010 |
| | 160168550 |
| SP-D | 160168450 |

# ANNEX 4. CODE FOR COMORBIDITY AND MEDICAL HISTORY

| Comorbidity / Medical history | Codes |
|-----------------------------------|--------|
| Coronary heart disease | 120-25 |
| Gastro-esophageal reflux disease | K21 |
| Obstructive sleep apnoea syndrome | G473 |
| COPD | J41-44 |
| Lung cancer | C34 |
| Pulmonary hypertension | 127 |

#### ANNEX 5. ALGORITHMS FOR DEFINING UDERLYING DISEASES

The following three subgroups will be defined to assess the distribution of underlying diseases and to perform subgroup analysis by underlying diseases.

Subgroup1: Autoimmune ILD, Non-autoimmune ILD, Multiple, Unknown, IPF#

Subgroup2: Hypersensitive pneumonitis, Exposure-related ILD, iNSIP, Unclassifiable IIP,

Sarcoidosis, RA-ILD, SSc-ILD, MCTD-ILD, Other autoimmune ILD, Other ILD, Multiple, Unknown, IPF<sup>#</sup>

Subgroup3: Hypersensitive pneumonitis, Exposure-related ILD, iNSIP, Unclassifiable IIP, Sarcoidosis, RA-ILD, SSc-ILD, MCTD-ILD, SLE-ILD, PM/DM-ILD, Sjogren ILD, Other autoimmune ILD, Other ILD, Multiple, Unknown, IPF#

#Note: Patients grouped into IPF are excluded from study population according to the exclusion criteria.

The patients will be grouped according to the following three steps.

Step 1: Patients will be grouped based on the fibrosing-ILD code on the index date

If two or more different (1) disease codes specified in this step 1 exist on index date

, then subgroup1=subgroup2=subgrou3=Multiple

**else if** disease code on index date=8844510, **then** Subrgoup1=Autoimmune ILD, subgroup2=SSc-ILD, subgroup3=SSc-ILD

**else if** disease code on index date=8847737, **then** subgroup1=Autoimmune ILD, subgroup2=RA-ILD, subgorup3=RA-ILD

**else if** disease code on index date=8848382, **then** subrgoup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=Other autoimmune ILD

else if disease code on index date=in(8848278, 8836513, 8844341), then subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD. Subgroup3=SLE-ILD

else if disease code on index date=in(8848267, 8848302, 8839362, 8848283, 8837013), then subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=PM/DM ILD else if disease code on index date=8834158, then subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=Sjogren ILD

(1)Note: The disease codes in the same conditional statement are NOT considered different. For example, disease codes of 8848278 and 8836513 are in the same conditional statement and these are not considered different disease codes. On the other hand, disease codes of 8848278 and 8848267 are in the different conditional statement and these are considered different disease codes.

Step 2: Patients not grouped in the step 1 will be grouped based on the earliest underlying disease code in the lookback period and fibrosing-ILD code on the index date

else if two or more different <sup>(2)</sup> earliest underlying disease codes specified in this step 2 exist AND disease code on index date=in(J84.1, J84.9), then subgroup1=subgroup2=subgrou3=Multiple else if earliest underlying disease code=in(D86.0, D86.1, D86.3, D86.8, D86.9) AND disease code on index date=in(J84.1, J84.9), then subgroup1=Non-autoimmune ILD, subgroup2=Sarcoidosis, subgroup3=Sarcoidosis

else if earliest underlying disease code=in(J67.0, J67.1, J67.2, J67.3, J67.4, J67.5, J67.6, J67.7, J67.8, J67.9) AND disease code on index date=in(J84.1, J84.9), then subgroup1=Non-autoimmune ILD, subgroup2=Hypersensitive pneumonitis, subgroup3=Hypersensitive pneumonitis else if earliest underlying disease code=J84.0 AND disease code on index date=in(J84.1, J84.9), then subgroup1=Non-autoimmune ILD, subgroup2=Other ILD, subgroup3=Other ILD else if earliest underlying disease code=in(J60, J61, J62.8, J63.0, J63.1, J63.2, J63.3, J63.4, J63.5, J64, J65, J66.0, J66.1, J68.0, J68.4, J70.1, J70.3, J70.4, J70.8) AND disease code on index date=in(J84.1, J84.9), then subgroup1=Non-autoimmune ILD, subgroup2=Exposure-related ILD, subgroup3=Exposure-related ILD

Note: Disease codes of 8840951 and 8848245 are added to the coitional statement.

else if earliest underlying disease code=in(M05.0, M05.1, M05.2, M05.3, M05.8, M05.9, M06.0, M06.2, M06.3, M06.4, M06.8, M06.9) AND disease code on index date=in(J84.1, J84.9, <u>8840951</u>, <u>8848245</u>), then subgroup1=Autoimmune ILD, subgroup2=RA-ILD, subgroup3=RA-ILD

else if earliest underlying disease code=in(M32.1, M32.9) AND disease code on index date=in(J84.1, J84.9, 8840951, 8848245), then subgroup1=Autoimmune ILD, subgroup2=Other

**else if** earliest underlying disease code=in(M33.0, M33.1, M33.2, M33.9) AND disease code on index date=in(J84.1, J84.9, <u>8840951</u>, <u>8848245</u>), **then** subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3= PM/DM ILD

autoimmune ILD, subgroup3=SLE-ILD

else if earliest underlying disease code=in(M34.0, M34.1, M34.8, M34.9) AND disease code on index date=in(J84.1, J84.9, <u>8840951</u>, <u>8848245</u>), then subgroup1=Autoimmune ILD, subgroup2=SSc-ILD, subgroup3=SSc-ILD

**else if** earliest underlying disease code=M35.0 AND disease code on index date=in(J84.1, J84.9, 8840951, 8848245), **then** subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=Sjogren ILD

**else if** earliest underlying disease code=7109008 AND disease code on index date=in(J84.1, J84.9, 8840951, 8848245), **then** subgroup1=Autoimmune ILD, subgroup2=MCTD-ILD, subgroup3=MCTD-ILD

**else if** earliest underlying disease code=in(8841317, 8850417, 8848245, M35.2, M35.3, M35.4, M35.5, M35.6, M35.7, M35.8, M35.9, M30.0, M30.1, M30.2, M30.3, M30.8, M31.0, M31.1, M31.2, M31.3, M31.4, M31.6, M31.7, M31.8, M31.9) AND disease code on index date=in(J84.1, J84.9, <u>8840951, 8848245</u>), **then** subgroup1= Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=Other autoimmune ILD

(2)Note: The earliest underlying disease codes in the same conditional statement are NOT considered different. For example, earliest underlying disease codes of D86.0 and D86.1 are in the same conditional statement and these are not considered different earliest underlying disease codes. On the other hand, earliest underlying disease codes of D86.0 and J67.0 are in the different conditional statement and these are considered different earliest underlying disease codes.

# Step 3: Patients not grouped in the step 1 and 2 will be grouped based on the fibrosing-ILD code on the index date

else if disease code on index date=in(5163005, 5150011, 8849927) AND no other fibrosing-ILD code on the index date, then subgroup1=subgroup2=subgroup3=IPF. These patients will be excluded from study population.

**else if** two or more different <sup>(3)</sup> disease codes including disease code of IPF specified in this step 3 exist on index date, **then** subgroup1=subgroup2=subgrou3=Multiple

else if disease code on index date=in(8850547, 8845727), then subgroup1=Non-autoimmune ILD, subgroup2=iNSIP, subgroup3=iNSIP

else if disease code on index date=in(5168008, 5168009, 5150001, 8845731, 8845640, J84.9), then subgroup1=Non-autoimmune ILD, subgroup2=Unclassifiable IIP, subgroup3=Unclassifiable IIP

else if disease code on index date=in(1363003, 8845663, 8845714, 8845719, 5168010), then subgroup1=Non-autoimmune ILD, subgroup2=Other ILD, subgroup3=Other ILD else if disease code on index date=in(8840951, 8848245), then subgroup1=Autoimmune ILD, subgroup2=Other autoimmune ILD, subgroup3=Other autoimmune ILD else subgroup1=subgroup2=subgroup3=Unknown

(3)Note: The disease codes in the same conditional statement are NOT considered different. For example, disease codes of 8850547 and 88457271 are in the same conditional statement and these are not considered different disease codes. On the other hand, disease codes of 8850547 and 5168008 are in the different conditional statement and these are considered different disease codes. **END** 

# ANNEX 6. INFORMATION OF THE CODE TO DEFINE FIBROSING ILD AND UNDERLYING DISEASES

| Disease | ICD-<br>10<br>Code | billing<br>code | Underlying<br>Autoimmune<br>Disease | ILD Category | Pre-Specified ILD<br>Clinical Diagnosis |
|---|---|---|---|---|---|
| respiratory disorder in dermatosclerosis | M348 | 8844510 | autoimmune | SSc-ILD | SSc-ILD |
| rheumatoid arthritis<br>interstitial pneumonia | M0510 | 8847737 | autoimmune | RA-ILD | RA-ILD |
| respiratory disorder<br>complicated by<br>granulomatosis with<br>polyangiitis | M313 | 8848382 | autoimmune | Other<br>autoimmune<br>ILDs | Other autoimmune ILDs |
| systemic lupus<br>erythematosus interstitial<br>pneumonia | M321 | 8848278 | autoimmune | SLE-ILD | other autoimmune<br>ILDs |
| respiratory disorder in systemic lupus erythematosus | M321 | 8836513 | autoimmune | SLE-ILD | other autoimmune<br>ILDs |
| interstitial pneumonia in juvenile dermatomyositis | M330 | 8848267 | autoimmune | PM/DM ILD | other autoimmune ILDs |
| interstitial pneumonia in dermatomyositis | M331 | 8848302 | autoimmune | PM/DM ILD | other autoimmune<br>ILDs |
| respiratory disorder in dermatomyositis | M331 | 8839362 | autoimmune | PM/DM ILD | other autoimmune<br>ILDs |
| interstitial pneumonia in polymyositis | M332 | 8848283 | autoimmune | PM/DM ILD | other autoimmune<br>ILDs |
| respiratory disorder in polymyositis | M332 | 8837013 | autoimmune | PM/DM ILD | other autoimmune ILDs |
| respiratory disorder in<br>Sjogren's syndrome | M350 | 8834158 | autoimmune | Sjogren ILD | other autoimmune ILDs |

| Disease | ICD-10<br>Code | billing<br>code | Underlying Autoimmune Disease | ILD<br>Category | Pre-Specified ILD Clinical Diagnosis |
|---|---|---|---|---|---|
| postinflammatory pulmonary fibrosis | J841 | 8845640 | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| usual interstitial pneumonia | J841 | 5168008 | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| idiopathic interstitial pneumonia | J841 | 5168009 | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| diffuse interstitial pneumonia | J841 | 5150001 | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| diffuse alveolar damage | J841 | 8845731 | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| idiopathic pulmonary fibrosis | J841 | 5163005 | IPF | IPF | IPF |
| pulmonary fibrosis | J841 | 5150011 | IPF | IPF | IPF |
| combined pulmonary fibrosis and emphysema | J841 | 8849927 | IPF | IPF | IPF |
| Idiopathic nonspecific interstitial pneumonia | J841 | 8850547 | Non-autoimmune | iNSIP | iNSIP |

| nonspecific interstitial pneumonia | J841 | 8845727 | Non-autoimmune | iNSIP | iNSIP |
|---|---|---|---|---|---|
| acute interstitial pneumonia | J84.1 | 1363003 | Non-autoimmune | Other IIPs | Other IIPs |
| respiratory bronchiolitis-associated interstitial lung disease | J841 | 8845663 | Non-autoimmune | Other IIPs | Other IIPs |
| cryptogenic organizing pneumonia | J841 | 8845714 | Non-autoimmune | Other IIPs | Other IIPs |
| desquamative interstitial pneumonia | J841 | 8845719 | Non-autoimmune | Other IIPs | Other IIPs |
| lymphocytic interstitial pneumonia | J841 | 5168010 | Non-autoimmune | Other IIPs | Other IIPs |
| - | - | - | Non-autoimmune | Unclassifiabl<br>e | Unclassifiable |
| interstitial pneumonia | J849 | 4860015 | Non-autoimmune | Unclassifiabl e | Unclassifiable |
| interstitial lung disease | J849 | 5168003 | Non-autoimmune | Unclassifiabl e | Unclassifiable |
| respiratory disorder in dermatosclerosis | M348 | 8844510 | | SSc-ILD | SSc-ILD |
| respiratory disorder complicated by granulomatosis with polyangiitis | M313 | 8848382 | | other CTD- | other CTD-ILD |
| lupus pneumonia | M321 | 8844341 | | SLE-ILD | SLE-ILD |

| systemic lupus erythematosus interstitial pneumonia | M321 | 8848278 | SLE-ILD | SLE-ILD |
|---|---|---|---|---|
| respiratory disorder in systemic lupus erythematosus | M321 | 8836513 | SLE-ILD | SLE-ILD |
| interstitial pneumonia in juvenile dermatomyositis | M330 | 8848267 | PM/DM-ILD | PM/DM-ILD |
| interstitial pneumonia in dermatomyositis | M331 | 8848302 | PM/DM-ILD | PM/DM-ILD |
| respiratory disorder in dermatomyositis | M331 | 8839362 | PM/DM-ILD | PM/DM-ILD |
| interstitial pneumonia in polymyositis | M332 | 8848283 | PM/DM-ILD | PM/DM-ILD |
| respiratory disorder in polymyositis | M332 | 8837013 | PM/DM-ILD | PM/DM-ILD |
| respiratory disorder in Sjogren's syndrome | M350 | 8834158 | Sjogren-ILD | Sjogren-ILD |
| interstitial pneumonia due to collagen disease | M351 | 8848245 | other CTD-<br>ILD | other CTD-ILD |
| rheumatoid lung disease | M0510 | 8840951 | other CTD-ILD | |
| rheumatoid arthritis interstitial pneumonia | M0510 | 8847737 | RA-ILD | RA-ILD |

N-Total number of study patients in each ILD underlying autoimmune disease category, IPF – Idiopathic Pulmonary Fibrosis, iNSIP – Idiopathic Nonspecific Interstitial Pneumonia, IIP – Idiopathic Interstitial Pneumonia, SSc-ILD – Systemic Sclerosis- Associated ILD, RA-ILD – Rheumatoid-Associated ILD, SLE-ILD – Systemic Lupus Erythematosus ILD, PM/DM ILD – Polymyositis/Dermatomyositis ILD

| Disease | ICD-<br>10<br>Code | billing code | Linkage Fibrotic code | Underlying<br>Autoimmune<br>Disease | ILD Category | Pre-Specified ILD<br>Clinical Diagnosis |
|---|---|---|---|---|---|---|
| Sjogren's syndrome | M350 | 7102001 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Sjogren ILD |
| Sjogren's syndrome<br>myopathy | M350 | 8841440 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Sjogren ILD |
| respiratory disorder in<br>Sjogren's syndrome | M350 | 8834158 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Sjogren ILD |
| primary Sjogren's<br>syndrome | M350 | 8848230 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Sjogren ILD |
| secondary Sjogren's<br>syndrome | M350 | 8848298 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Sjogren ILD |

| overlap syndrome | M351 | 8841317 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
|---|---|---|---|---|---|---|
| anti-ARS antibody<br>syndrome | M351 | 8850417 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| mixed connective tissue disease | M351 | 7109008 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | MCTD-ILD | MCTD-ILD |
| interstitial pneumonia<br>due to collagen<br>disease | M351 | 8848245 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| Behcet's disease | M352 | 1361002 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| vulval Behcet's<br>disease | M352 | 1361011 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |

| ocular Behcet's<br>disease | M352 | 8845881 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
|---|---|---|---|---|---|---|
| vasculo-Behcet's<br>disease | M352 | 1361009 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| oral Behcet's disease | M352 | 1361010 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| neuro-Behcet disease | M352 | 1361005 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| entero-Behcet<br>disease | M352 | 8842203 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| incomplete Behcet disease | M352 | 8846052 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| polymyalgia<br>rheumatica | M353 | 7250004 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |

| diffuse eosinophilic<br>fasciitis | M354 | 8839540 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
|---|---|---|---|---|---|---|
| eosinophilic fasciitis | M354 | 7294009 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| acrosclerosis | M355 | 7108005 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| multifocal<br>fibrosclerosis | M355 | 8836987 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| Weber-Christian disease | M356 | 8830767 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| hyperkinetic<br>syndrome | M357 | 7285007 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |

| familial ligament relaxation | M357 | 8831279 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
|---|---|---|---|---|---|---|
| eosinophilia-myalgia<br>syndrome | M358 | 7101038 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| IgG4-related disease | M359 | 8848113 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| systemic autoimmune<br>disease | M359 | 8836526 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| collagen disease | M359 | 7109004 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| anemia associated<br>with collagen<br>disease | M359 | 8833428 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| pericarditis of collagen disease | M359 | 4239017 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmune/CTD<br>ILD | Other-<br>autoimmune/CTD<br>ILD |
| polyarteritis nodosa | M300 | 8833125 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |

| eosinophilic<br>granulomatosis with<br>polyangiitis | M301 | 8848338 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
|---|---|---|---|---|---|---|
| juvenile multiple<br>arteritis | M302 | 8835258 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| acute febrile<br>mucocutaneous<br>lymph node<br>syndrome | M303 | 4461009 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| Kawasaki's disease | M303 | 4461003 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| ischemic heart<br>disease due to<br>Kawasaki's disease | M303 | 8831474 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| Kawasaki disease-<br>related coronary<br>artery aneurysm | M303 | 4461004 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| incomplete Kawasaki<br>disease | M303 | 8846336 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| polyangiitis overlap<br>syndrome | M308 | 8837016 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |

| skin polyarteritis<br>nodosa | M308 | 8846209 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
|---|---|---|---|---|---|---|
| cutaneous arteritis | M308 | 8849445 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD | Other-<br>autoimmue/CTD<br>ILD |
| Goodpasture's syndrome | M310 | 4462001 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| hypersensitivity vasculitis | M310 | 4462002 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| cutaneous<br>leukocytoclastic<br>vasculitis | M310 | 8851019 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| drug-induced<br>hypersensitivity<br>vasculitis | M310 | 8844108 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| thrombotic<br>thrombocytopenic<br>purpura | M311 | 4466002 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| thrombotic<br>microangiopathy | M311 | 8833136 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| acquired thrombotic<br>thrombocytopenic<br>purpura | M311 | 8849965 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| congenital thrombotic<br>thrombocytopenic<br>purpura | M311 | 8847881 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| gangrenous rhinitis | M312 | 4609006 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |

| localized<br>granulomatosis with<br>polyangiitis | M313 | 8848336 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
|---|---|---|---|---|---|---|
| generalized<br>granulomatosis with<br>polyangiitis | M313 | 8848371 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| granulomatosis with polyangiitis | M313 | 8848381 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| respiratory disorder<br>complicated by<br>granulomatosis with<br>polyangiitis | M313 | 8848382 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| Takayasu's arteritis | M314 | 8848380 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| aortitis syndrome | M314 | 4467003 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| - | - | - | - | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| giant cell arteritis | M316 | 4465001 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |

| microscopic<br>polyangiitis | M317 | 8842086 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
|---|---|---|---|---|---|---|
| ANCA-associated vasculitis | M318 | 8845513 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| hypocomplementemic urticarial vasculitis | M318 | 8849413 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| necrotizing angitis | M319 | 4460015 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |
| polyangiitis | M319 | 4460017 | J84.1, J84.8, J84.9,<br>J99.0, J99.1 | Autoimmune | Other-<br>autoimmue/CTD<br>ILD | Other-<br>autoimmue/CTD<br>ILD |

N-Total number of study patients in each ILD underlying autoimmune disease category,
SSc-ILD – Systemic Sclerosis- Associated ILD, RA-ILD – Rheumatoid-Associated ILD, SLE-ILD – Systemic Lupus Erythematosus ILD, PM/DM ILD –
Polymyositis/Dermatomyositis ILD

CTD-ILD – connective tissue disease- associated ILD, MCTD-ILD – Mixed Connective Tissue Disease-ILD

#### **ANNEX 7. REVIEWERS AND APPROVAL SIGNATURES**

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | Х | Х |
| Global TM Epi | X | Х | Х |
| Global TMM / TMMA / TM Market Access | Х | Х | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | Х | Х |
| Global CTIS representative | Х | | |
| Local Medical Director | X (if local study) | | Х |
| Local Head MAcc / HEOR Director | X (if local study) | | Х |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical Development<br>/ Medical Affairs / Market Access* | Х | Х | |
| Global TA Head PV RM* | X | | |
| RWE CoE | Х | Х | |
| PSTAT / PSTAT-MA (for NISnd only) | Х | Х | Х |
| NIS DM | X | Х | Х |
| Local Head MA/Clinical Development | | | X (does not apply to NISed without chart abstraction) |

<sup>\*</sup> After review by Global TM for function

## Study Title:

lincidence probability of progression to progressive fibrosing interstitial lung diseases (PF-ILDs) in non-IPF fibrosing ILD patients and their current management and treatments in Japan **Study Number**:

#### **Protocol Version:**

Version 1.2

## **BOEHRINGER INGELHEIM Group of Companies**

**NIS Protocol Template** 

Study number: <insert> Document number: <insert>

I herewith certify that I agree to the content of the study protocol and to all documents referenced in the study protocol.

| Position: PI_ | Name/Date: <b>N/A</b> | Signature: |
|--------------------------------|-----------------------|----------------|
| Position: NIS | Name/Date: | |
| Position: <u>Japan Med</u> | Name/Date: | Signature: |
| Position: <u>Global TM Epi</u> | Name/Date: | Signature: |
| Position: | Name/Date: | <br>Signature: |
| Position: | Name/Date: | <br>Signature: |
| Position: | Name/Date: | <br>Signature: |

Page 41 of 41